CLINICAL TRIAL: NCT04720274
Title: Utilizing EMG Shorts to Access Hip Injuries and Recovery After Surgery
Brief Title: Utilizing EMG Shorts in Hip Population
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator decided to not open the study.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00104994
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Hip Injuries
Keywords: EMG Shorts; Hip Pain
MeSH Terms: conditions — Hip Injuries | interventions — Electromyography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Participants with Hip Pain or Injuries (Experimental)
  Interventions: Device: Electromyopathy (EMG) Shorts
- Healthy Participants (Active Comparator)
  Interventions: Device: Electromyopathy (EMG) Shorts

INTERVENTIONS:
Device: Electromyopathy (EMG) Shorts — Participants will be asked to complete physical activities while wearing EMG shorts

SUMMARY:
The purpose of this study is to use a combination of electromyopathy (EMG) shorts and muscle monitoring software to collect data from participants performing physical exercises in order to determine the combination's diagnostic efficacy and ability to provide rehabilitative guidance for people who are recovering from hip injuries. Both healthy volunteers and Duke Patients seeking treatment for their hip pain and/or injuries will be enrolled in our research. If participants choose to take part they will be asked to wear these EMG shorts and perform various exercises like running on a treadmill, riding a stationary bike, or lifting weights.

Participation in this study consists of one study visit for healthy volunteers, but will last up to six months for Duke Patients. At each standard of care clinic visit throughout six months, Duke Patients will be asked to also come in for a study visit, wear the EMG shorts, and perform the same exercises preformed during the first study visit.

ELIGIBILITY:
Inclusion Criteria:

Inclusion (Duke Patients):

* All subjects must be 18 years of age or older.
* Any patient that currently has hip pain or injury and is seeking treatment from either Dr. Mather, Dr. Lewis, or Dr. Olson, within the hip preservation clinics.
* Subjects must be able to fit into the shorts in order to participate.

Inclusion (Healthy Volunteers):

* All healthy volunteer subjects must be 18 years of age or older.
* Subjects must be able to fit into the shorts in order to participate.

Exclusion Criteria:

Exclusion (Duke Patients):

* Any recent lower extremity injury (such as an ankle sprain/surgery or knee surgery).
* Patient is unable to provide written consent, or patient is unable to speak, write, or understand English.
* Pregnant women (Verbal Confirmation)
* Allergic or hypersensitivity to laminate material.

Exclusion (Healthy Volunteers):

* Any recent lower extremity injury (such as an ankle sprain/surgery or knee surgery).
* Prior hip surgery, or current hip injury, surgery, or pain.
* Patient is unable to provide written consent, or patient is unable to speak, write, or understand English.
* Pregnant women (Verbal Confirmation)
* Allergic or hypersensitivity to laminate material.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-04 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Amount of muscle activation while preforming physical therapy exercises in a post operative setting as measured EMG shorts. | Up to 6 months

SECONDARY OUTCOMES:
Percent of participants that stated a positive experience with EMG shorts as measured by patient satisfaction survey. | End of study, up to one year
  Study team developed survey, one to two question survey about experience.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Mather, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No